CLINICAL TRIAL: NCT03362788
Title: Contemporary Antithrombotic Treatment in Patients With Non-valvular AF Undergoing PCI: The Greek AntiPlatElet Atrial Fibrillation (GRAPE-AF) Registry.
Brief Title: The Greek AntiPlatElet Atrial Fibrillation Registry.
Acronym: GRAPE-AF
Status: Completed | Type: Observational
Sponsor: Attikon Hospital (Other)
Collaborators: Hellenic Cardiology Society (Other)
Responsible Party: Principal Investigator, Dimitrios Alexopoulos, Professor of Cardiology, Attikon Hospital
Other Study IDs: AttikonHGR
Record Dates: First submitted 2017-11-24; First posted 2017-12-05 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Atrial Fibrillation; Coronary Artery Disease
Keywords: Antithrombotics Antiplatelets Stents Angioplasty
MeSH Terms: conditions — Atrial Fibrillation; Coronary Artery Disease | interventions — acarboxyprothrombin; N(4)-oleylcytosine arabinoside

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- VKA: Patients receiving VKA as anticoagulant treatment plus a P2Y12 inhibitor (clopidogrel 75mg or ticagrelor 90mg twice daily) and/or aspirin ≤100mg daily.
  Treatment will be at operator's discretion or, post discharge, at prescribing physician's discretion.
  Interventions: Drug: VKA
- NOAC: Patients receiving a NOAC as anticoagulant treatment plus a P2Y12 inhibitor (clopidogrel 75mg or ticagrelor 90mg twice daily) and/or aspirin ≤100mg daily.
  Treatment will be at operator's discretion or, post discharge, at prescribing physician's discretion.
  Interventions: Drug: NOAC

INTERVENTIONS:
Drug: VKA — VKA plus a P2Y12 inhibitor (clopidogrel 75mg or ticagrelor 90mg twice daily) and/or aspirin ≤100mg daily.
  Other Names: Vitamin K antagonist
  Groups: VKA
Drug: NOAC — NOAC plus a P2Y12 inhibitor (clopidogrel 75mg or ticagrelor 90mg twice daily) and/or aspirin ≤100mg daily.
  Other Names: Non-vitamin K oral anticoagulant
  Groups: NOAC

SUMMARY:
Approximately 5% to 7% of patients undergoing percutaneous coronary intervention for the treatment of coronary artery disease, require chronic oral anticoagulation on top of aspirin and a P2Y12 receptor antagonist, mainly due to non-valvular atrial fibrillation. Advent of non-vitamin K antagonist oral anticoagulants (NOAC) increased treatment options, while there is cumulative evidence that dual combination of NOAC and P2Y12 receptor antagonist attenuates bleeding without compromising efficacy. Greek AntiPlatElet Atrial Fibrillation (GRAPE-AF) is an observational study of non-valvular atrial fibrillation patients undergoing percutaneous coronary intervention, planning to enroll >500 participants during 1 year period in Greece. Patients will be followed-up at 1, 6 and 12 months post hospital discharge. Key data to be collected pre-discharge include demographics, detailed past medical history, antithrombotic and concomitant treatment. Study's primary endpoint is clinically significant bleeding defined as Bleeding Academic Research Consortium (BARC) ≥2) at 12 months, between vitamin K antagonists (VKAs) and NOACs-treated patients. All clinical events will be adjudicated by an independent endpoint committee.This study would provide "real world" information on current antithrombotic treatment patterns and clinical outcome of patients with non-valvular atrial fibrillation undergoing percutaneous coronary intervention.

DETAILED DESCRIPTION:
All consecutive patients undergoing percutaneous coronary intervention over 1 year period will be screened for participation. Discharge antithrombotic medication will be at the discretion of the treating physician.

Follow-up visits will be performed at 1, 6 and 12 months post-percutaneous coronary intervention by telephone contact or personal interview. All outcome and adverse events will be adjudicated by an independent endpoint committee. All data will be recorded in electronic forms and multiple quality controls will be performed both electronically and on-site to ensure data integrity.

Platelet reactivity substudy:Patients receiving either clopidogrel or ticagrelor as part of their (dual or triple) combination therapy, will be eligible for sub-study of platelet function assessment with the VerifyNow assay at 1 month post-percutaneous coronary intervention in centers with test availability.

Sub-study's endpoints will be platelet reactivity between groups and high platelet reactivity rate between groups.

ELIGIBILITY:
Inclusion Criteria:

Percutaneous coronary intervention with stent implantation Non-valvular atrial fibrillation (paroxysmal, persistent or permanent) with indication for anticoagulation Written informed consent

Exclusion Criteria:

1. Any clinically significant bleeding (BARC ≥2) at the time of screening or within the previous month
2. Prior intracranial bleeding
3. Dialysis or calculated creatinine clearance <30 mL/min at screening
4. Known significant liver disease (eg, acute hepatitis, chronic active hepatitis, cirrhosis), or liver function test abnormalities at screening (confirmed with repeat testing): alanine transaminase (ALT) >5 times the upper limit of normal or ALT >3 times the upper limit of normal plus total bilirubin >2 times the upper limit of normal
5. A PT or INR test result that is higher than the upper limit of normal at the time of screening that suggests an underlying coagulation disorder (except for subjects taking VKA), or an INR that does not drop to 2.5 or below by 72 h after sheath removal following the index procedure.
6. Life expectancy of less than 12 months
7. Incomplete staged percutaneous coronary intervention procedure (once the completion of the staged procedure has occurred, the final percutaneous coronary intervention PCI may become the index event and is allowed)
8. Planned coronary artery bypass grafting
9. Contraindications to the use of clopidogrel or ticagrelor or NOAC, per prescribing information (e.gHypersensitivity to the active substance or to any of the excipients or co-administration with strong CYP3A4 inhibitors e.g. ketoconazole, clarithromycin, nefazodone, ritonavir, and atazanavir).
10. Estimated high risk of non-availability for follow-up visits

Ages: 20 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All consecutive patients undergoing percutaneous coronary intervention over 1 year period will be screened for atrial fibrillation and need for anticoagulation plus P2Y12 receptor antagonist.
Sampling Method: Probability Sample
Enrollment: 654 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Clinically significant bleeding | 12 months
  Clinically significant bleeding defined as Bleeding Academic Research Consortium (BARC) ≥2 between the 2 groups (VKA vs NOACs).

SECONDARY OUTCOMES:
MACEs | 12 months
  MACEs (cardiovascular death, ischemic stroke, myocardial infarction, systemic embolism and unplanned coronary revascularization) between the 2 groups (VKA vs NOACs)
Net clinical endpoint | 12 months
  Net clinical endpoint includes cardiovascular death, ischemic stroke, myocardial infarction, systemic embolism, unplanned coronary revascularization and BARC ≥2 bleedings between the 2 groups (VKA vs NOACs)

OTHER OUTCOMES:
HAS-BLED score | 12 months
  Validation of baseline HAS-BLED score (between 0 and 9) in predicting bleeding events and evaluation of their impact on antithrombotic medication at discharge. Higher values represent a worse outcome.
CHA2DS2-VASc Score | 12 months
  Validation of CHA2DS2-VASc Score (between 0 and 9) in predicting ischemic stroke and evaluation of its impact on antithrombotic medication at discharge.Higher values represent a worse outcome.
Charlson Comorbidity Index (CCI) | 12 months
  Validation of Charlson Comorbidity Index (CCI) in predicting bleeding events and ischemic stroke and evaluation of its impact on antithrombotic medication at discharge.
Anticoagulation and Risk Factors In Atrial Fibrillation (ATRIA) score | 12 months
  Validation of ATRIA score (0 to 15) in predicting bleeding events and evaluation of their impact on antithrombotic medication at discharge. Higher values represent a worse outcome.
Outcomes Registry for Better Informed Treatment of Atrial Fibrillation (ORBIT) score | 12 months
  Validation of ORBIT score (0 to 7) in predicting bleeding events and evaluation of their impact on antithrombotic medication at discharge.Higher values represent a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Alexopoulos, MD, Principal Investigator — Attikon Hospital
Locations (1):
- Attikon University Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Alexopoulos D, Dragona VM, Varlamos C, Ktenas D, Lianos I, Patsilinakos S, Sionis D, Zarifis I, Bampali T, Poulimenos L, Skalidis E, Pissimisis E, Trikas A, Tsiafoutis I, Kafkas N, Olympios C, Tziakas D, Ziakas A, Voudris V, Kanakakis I, Tsioufis C, Davlouros P, Benetou DR. One-Year Outcomes in Anticoagulated Atrial Fibrillation Patients Undergoing Percutaneous Coronary Intervention: Insights From the Greek Antiplatelet Atrial Fibrillation Registry. J Cardiovasc Pharmacol. 2023 Feb 1;81(2):141-149. doi: 10.1097/FJC.0000000000001389. PMID 36410034
- [Derived] Benetou DR, Varlamos C, Ktenas D, Tsiafoutis I, Koutouzis M, Bampali T, Mantis C, Zarifis J, Skalidis E, Aravantinos D, Varvarousis D, Lianos I, Kanakakis J, Pisimisis E, Ziakas A, Davlouros P, Alexopoulos D; GRAPE-AF investigators. Trends of Antithrombotic Treatment in Atrial Fibrillation Patients Undergoing Percutaneous Coronary Intervention: Insights from the GReek-AntiPlatElet Atrial Fibrillation (GRAPE-AF) Registry. Cardiovasc Drugs Ther. 2021 Feb;35(1):11-20. doi: 10.1007/s10557-020-07090-x. Epub 2020 Oct 9. PMID 33034806